CLINICAL TRIAL: NCT06070935
Title: Nailfold Capillaroscopic Assessment in Pediatric Uveitis Patients
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Maha Sayed Ibrahim Abdelrahman, Principal invesigator, Assiut University
Other Study IDs: Nailfold capillaroscopy
Record Dates: First submitted 2023-10-01; First posted 2023-10-06 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Uveitis
MeSH Terms: conditions — Uveitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- pediatric uveitis: pediatric uveitis patients < 18 years old
- healthy subjects: healthy subjects< 18 years old

SUMMARY:
Pediatric uveitis accounts for 5-10% of uveitis cases. it may be infectious or noninfectious in etiology. The etiology of noninfectious uveitis may be autoimmune. The most common causes of pediatric uveitis are idiopathic and juvenile idiopathic arthritis-associated uveitis. Uveitis morbidities in pediatric patients include cataract, glaucoma, and amblyopia. Pediatric uveitis may be accopanied by involvement of the ocular vasculature, such as retinal vasculitis. We hypothesize that there are differences in systemic microcirculation between pediatric uveitis patients and healthy pediatric controls.

DETAILED DESCRIPTION:
The systemic microcirculation will be investigated through nailfold capillaroscopic (NFC) assessment with noninfectious uveitis and healthy pediatric controls.

The NFC parameters are:

capillary density (number of capillaries per mm), dilated capillaries (apex of >20µm), avascular areas, the presence of microhemorrhages, and capillary morphology (normal, multiple crossings, tortuous, bushy, ramified, non-convex, or bizarre capillaries).

ELIGIBILITY:
Inclusion Criteria:

* patients with uveitis < 18 years old

Exclusion Criteria:

* infectious uveitis
* age > 18 years old

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: pediatric uveitis patients and healthy pediatric control
Sampling Method: Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
capillary density by nailfold capillaroscopy | 6 months
  (number of capillaries per mm)
detection of number of dilated capillaries by nailfold capillaroscopy | 6 months
  number of dilated capillaries (apex of >20µm)
detection of other abnormalities as avascular areas, microhemorrhages, and abnormal capillary morphology | 6 months
  detection of multiple crossings, tortuous, bushy, ramified, non-convex, or bizarre capillaries

SECONDARY OUTCOMES:
correlation of nailfold findings with uveitis activity | 6 months
  correlation of capillary abnormalities detected with active uveitis.

CONTACTS AND LOCATIONS:
Overall Officials: Maha Abdelrahman, MD, PHD, Principal Investigator — Assiut University
Locations (1):
- Maha Abdelrahman, Asyut, Egypt